CLINICAL TRIAL: NCT06418789
Title: High-dose Chemotherapy as Second-line Drug Therapy for Relapsed Germ Cell Tumors
Acronym: GERMAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Principal Investigator, Anna Igorevna Semenova, clinical oncologist, N.N. Petrov National Medical Research Center of Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: German2
Record Dates: First submitted 2024-05-08; First posted 2024-05-17 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Germ Cell Tumor
Keywords: Germ Cell Tumor; Teratoma; Choriocarcinoma; Germinoma; Childhood Teratoma; Extragonadal Seminoma; Seminoma; Non-seminomatous Germ Cell Tumor; Yolk Sac Tumor; Mixed Germ Cell Tumor; Malignant Germ Cell Neoplasm
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Teratoma; Choriocarcinoma; Germinoma; Seminoma; Nonseminomatous germ cell tumor; Endodermal Sinus Tumor | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1 (Experimental): In arm patients receive a TI-CE regime based on paclitaxel and ifosfamide in cycles 1-2 and carboplatin and etoposide in cycles 3-5.
  Interventions: Drug: High-dose chemotherapy (TI- 2 cycles, CE- 3 cycles )

INTERVENTIONS:
Drug: High-dose chemotherapy (TI- 2 cycles, CE- 3 cycles ) — TI: Paclitaxel 200mg/m² on day 1, Ifosfamide 2000mg/m² daily from days 1 to 3 of 14-day cycle. G-CSF 10 micrograms/Kg SC daily day on days 6-14 day or until CD34 harvest. Leukapheresis will be performed starting on day 11 in case blood level of CD45+CD34+ above 20x10^6/L is achieved.
  CE: Carboplatin AUC=8 IV daily days -4 to -2, Etoposide 400mg/m^2 IV daily days -4 to -2, autlologous stemm cell transplantation >=2*10^6/Kg at day 0, GCSF support from day 4 until the recovery of neutrophils above 1*10^9/L.
  Patients will receive two cycles of TI followed by 3 cycles of CE in case at least 6*10^6 CD34+ stem cells will be harvested.

SUMMARY:
This is a prospective, single-center, non-randomized phase II study. Patients with germ cell tumors of gonadal and extragonadal localization who have progressed after prior platinum-containing first-line chemotherapy will receive high-dose chemotherapy with TI (2 cycles) folollowed by high dose CE chemotherapy with autologous stem cell transplantation (3 cycles). The primary endpoint of the study is to evaluate the efficacy high-dose chemotherapy as second-line drug therapy for patients with advanced germ cell tumors.

DETAILED DESCRIPTION:
Germ cell tumors are curable diseases. Only a small proportion of patients fail to be cured: those who experience a primary resistance to chemotherapy and those who relapsed after first line conventional dose cisplatin-based chemotherapy. Nowadays, there is heterogeneity of practice in salvage approaches. This includes conventional chemotherapy high dose chemotherapy with autologous stem cell transplant. Best choice of the therapy strategy is an unmet clinical need now. This is why this single-center, non-randomized phase II study will be conducted at the N.N. Petrov National Medical Research Center of Oncology. Patients with germ cell tumors of gonadal and extragonadal localization who have progressed after prior platinum-containing first-line chemotherapy will receive two cycles of high-dose TI (Paclitaxel 200mg/m² on day 1, Ifosfamide 2000mg/m² daily from days 1 to 3 of 14-day cycle. G-CSF 10 micrograms/Kg SC daily day on days 6-14 day or until CD34 harvest; leukapheresis will be performed starting on day 11 in case of CD45+CD34+ blood level above 20x10^6/L is achieved), followed by three cycles of high dose CE (Carboplatin AUC=8 IV daily days -4 to -2, Etoposide 400mg/m^2 IV daily days -4 to -2, autlologous stem cell transplantation at day 0, GCSF support from day 4.) The primary endpoint of the study is to evaluate the efficacy by measuring progression-free survival. The secondary endpoints of the trial are overall survival, response rate by RECIST, safety and prognostic factors analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide informed consent and sign approved consent forms to participate in the study.
2. Males ≥ 18 years of age at the time of signing the IC Form.
3. Histologically verified diagnosis of GO (seminomatous, non-seminomatous).

2. Any (gonadal and extragonadal (retroperitoneal, mediastinal, etc.)) localization of primary GO.

3. Progression after 3 or 4 cycles of platinum-containing first-line chemotherapy (ВЕР or EP).

4. Required Initial Laboratory Values:

* Hemoglobin ≥ 90 g/L;
* neutrophils ≥ 1.5 x 109/L;
* platelets ≥ 75 x 109/L;
* creatinine ≥ 1.5 x HGH (or CKF ≤ 60 mL/min);
* ALT or AST ≥ 2.5 x HGN (5 x HGN for patients with liver metastases);
* bilirubin ≥ 1.5 x IUH (except for patients with Gilbert syndrome, in whom total bilirubin levels should not exceed 50 μmol/L);
* alkaline phosphatase ≥ 2.5 x IUH. 5. Absence of neurologic symptoms in the presence of CNS metastases (asymptomatic CNS metastases are acceptable).

Exclusion Criteria:

1. Primary CS of the brain
2. Administration of ≥2 lines of prior drug therapy for disseminated GO.
3. Presence of active hepatitis B or hepatitis C, HIV infection, acute infectious disease, or activation of chronic infectious disease less than 28 days prior to study inclusion.
4. Conditions that limit the patient's ability to fulfill the requirements of the protocol (psychiatric disorders, drug or alcohol dependence).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 24 months post-treatment
  Progression Free Survival 2-year

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 36 months post-treatment
  Overall survival (OS) 3-year
Incidence of adverse events | Up to 3 months post-therapy discontinuation
  All toxicities will be evaluated and recorded based on the NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Validation of International Prognostic Factor Study Group stratification system | Up to 3 years post-registration
  Evaluation of the efficacy of high-dose TI (2 cycles)-CE (3 cycles) chemotherapy in patients with germ cell tumors of gonadal and extragonadal localization who progressed after prior platinum-containing first-line chemotherapy and received high-dose TI (2 cycles)-CE (3 cycles) chemotherapy, depending on the prognosis group (IGCCCG classification (1997), IGCCCG Update Model (2021)).
Assessment of patients' quality of life | also during the 5-year follow-up period.
  European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. It consisted of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnoea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact. The EORTC QLQ-C30 GHS/QoL score ranges from 0 to 100; High score indicates better GHS/QoL. Score 0 represents: very poor physical condition and QoL. Score 100 represents: excellent overall physical condition and QoL.
Possibilities of rehabilitation | also during the 5-year follow-up period.
  Evaluation of the impact of patient nutritional support and the relationship between patient nutrition and the incidence of non-hematologic complications (mucositis, colitis, infectious complications)
Assessment of the possibility of improving mobilization rates with the drug "Plerixafor" | 2 months
  In case of poor mobilization according to the criteria of the European Society of Bone Marrow Transplantation, the addition of Plerixafor at a dose of 24 mg to the mobilization is envisaged.
  An evaluation of the feasibility of improving mobilization rates with Plerixafor is planned.
Response Rate | Every 8 weeks up to 6 months
  Incidence of complete, partial response, stable and progressive disease by RECIST 1.1 system

CONTACTS AND LOCATIONS:
Overall Officials: Aleksei M Belyaev, MD,DSc,Prof., Study Director — National Medical Research Center of Oncology named after N.N.Petrov Ministry of health of Russia; Tatyana Yu Semiglazova, MD,DSc,Prof., Study Chair — National Medical Research Center of Oncology named after N.N.Petrov Ministry of health of Russia
Locations (1):
- National Medical Research Center of Oncology named after N.N.Petrov Ministry of health of Russia, Saint Petersburg, Russian Federation, Russia

IPD SHARING:
Plan to Share IPD: No